CLINICAL TRIAL: NCT03817528
Title: ITI-007 (Lumateperone Tosylate) for Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: ITI-007 approved by FDA
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey A. Lieberman, MD, Director, New York State Psychiatric Institute, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7716
Record Dates: First submitted 2018-11-30; First posted 2019-01-25 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — lumateperone

STUDY DESIGN:
Intervention Model Description: open-label
Masking Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ITI-007 (Experimental): Open-Label ITI-007 40-60 mg
  Interventions: Drug: ITI-007

INTERVENTIONS:
Drug: ITI-007 — ITI-007 (Lumateperone tosylate)dosed 40-60 mg based on efficacy/adverse events
  Other Names: Lumateperone tosylate

SUMMARY:
The purpose of this study is to offer open label ITI-007 treatment to patients who poorly respond or poorly tolerate approved medications.

DETAILED DESCRIPTION:
Patients will be started on ITI-007 and current medication will be slowly discontinued within the first 7 days of starting ITI-007, with some flexibility allowed if clinically indicated. No patients will be left unmedicated because of this study.

Patients will be seen weekly for the first 4 weeks, biweekly for the second month and then monthly for six months. Patients will be monitored by clinical and safety rating scales, and will be required to show improvement after 3 months to remain in this study. Patients not improving at this time will be assessed for the risks/benefits of continuing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) diagnosis of schizophrenia or schizoaffective disorder
* Has capacity to provide informed consent
* Medically stable for study participation
* Judged clinically not to be at significant suicide or violence risk
* Inadequate response or tolerability to previously antipsychotic therapy, as defined by at least one of the following: prior clozapine failure, a PANSS>80 despite at least six weeks of a current antipsychotic therapy, a Clinical Global Impressions scale-Improvement (CGI-I) of 4 after at least two six week trials of antipsychotics (retrospective assessment) or failure to tolerate an adequate dose of at least antipsychotics (as defined by the Physicians Desk Reference)

Exclusion Criteria:

* Substance abuse within last 90 days
* ECG abnormality that is clinically significant
* Pregnancy, lactation, or lack of use of effective birth control
* Presence or positive history of significant unstable medical or neurological illness (including any history of seizure disorder, hepatitis, renal insufficiency or mental retardation), history of HIV
* Clinically significant abnormal laboratory tests, positive for hepatitis B or C or liver function tests (LFTs) > 2x Upper Limit of Normal, use of strong CYP3A4 inhibitors or inducers
* History or presence of concomitant major psychiatric illness.
* Use of other antipsychotic medications at baseline.
* Use of another investigational medication in the previous 4 weeks

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Lieberman, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment reflects the number of participants were deemed eligible and received study drug
Pre-assignment Details: Participants underwent a screening phase to determine eligibility to receive study medication
Period: Overall Study
Arm/Group | ITI-007
Started | 4
Completed | 1
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Baseline population is participants who received at least one dose of study drug
Arm/Group | ITI-007
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Schizophrenia Symptoms
Description: schizophrenia symptoms will be measures using the Positive and Negative Symptom Scale (PANSS) Total PANSS score (range: 30-210). Individual items scored from 1(absent) to 7 (extremely severe). Total PANSS score is sum of the 30 individual items with lowest score (30) indicating all symptoms absent and the maximum score (210) indicating all symptoms rated as extremely severe.
Time Frame: Change from baseline in Total PANSS score after 6 month treatment
Population: Completed participants (6 months of treatment). Outcome measure reported as change in PANSS score from baseline to end of treatment
Measure: Number; unit: change in PANSS score from baseline
Arm/Group | ITI-007
Number analyzed (Participants) | 1
change in PANSS score from baseline | 11

ADVERSE EVENTS:
Time Frame: Adverse events to be reported from time of consent (whether received study drug or not) to 30 days after completion of study treatment (up to 8 months)
Description: AE/SAE collection from all individuals who signed informed consent (total: 8)
Arm/Group | ITI-007
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITI-007 (N=8)
worsening of symptoms (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITI-007 (N=8)
hypomania (Psychiatric disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT03817528/Prot_000.pdf